CLINICAL TRIAL: NCT01346046
Title: An Evaluation of a Noninvasive Diabetes Screening Device in Subjects at the TCOYD Diabetes Conference
Brief Title: Evaluation of SCOUT DS in Subjects With Type 2 Diabetes #2
Acronym: TCOYD2
Status: Completed | Type: Observational
Sponsor: VeraLight, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VL-2717
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes Mellitus, Non-Insulin Dependent
Keywords: Type 2 Diabetes; Adults 18 years and older; Taking Control of Your Diabetes Health Fair
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Those with Type 2 diabetes: 270 subjects with Type 2 diabetes
- Non diabetic: 30 healthy subjects

SUMMARY:
The primary objective of the trial is to collect SCOUT DS and Hemoglobin A1c measurements of subjects who have been diagnosed with Type 2 diabetes.

DETAILED DESCRIPTION:
Previous studies have excluded subjects with Type 2 diabetes. The primary objective of this study is to correct an imbalance in the disease prevalence of the data set used to develop the SCOUT DS diabetes screening algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years Self-reported diagnosis of type 2 diabetes No Self-reported diagnosis of type 2 diabetes

Exclusion Criteria:

* Less than 18 years of age

  * Diagnosed with type 1 diabetes
  * Known to be pregnant (Self Reported)
  * Receiving dialysis or having known renal compromise
  * Scars, tattoos, rashes or other disruption/discoloration on the left volar forearm.
  * Known to have, or at risk for, photosensitivity reactions ( e.g., sensitive to ultraviolet light, or taking medication known to cause photosensitivity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Attendees of the Taking Control of Your Diabetes Health Fair, Albuquerque Convention Center
Sampling Method: Non-Probability Sample
Enrollment: 264 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Continuing validation of SCOUT DS algorithm | 1 day
  Collect SCOUT DS and Hemoglobin A1c measurements of subjects with Type 2 Diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Walter Forman, MD, Principal Investigator — Lovelace Scientific Resources
Locations (1):
- Albuquerque Convention Center, Albuquerque, New Mexico, United States